CLINICAL TRIAL: NCT02588755
Title: Anti-tumor Recurrence With Transarterial Chemoembolization (TACE) Plus Tegafur Versus TACE on Patients With Intrahepatic Cholangiocarcinoma After Curative Resection：A Randomized Controlled Study
Brief Title: TACE Plus Tegafur Versus TACE for Intrahepatic Cholangiocarcinoma After Curative Resection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, ShenFeng, vice president of the Eastern Hepatobiliary Surgery Hospital, Eastern Hepatobiliary Surgery Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EHBHKY2015-0123
Record Dates: First submitted 2015-10-27; First posted 2015-10-28 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Intrahepatic Cholangiocarcinoma
Keywords: Chemoembolization; Therapeutic; Tegafur
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TACE+ Tegafur (Active Comparator): Patients will be treated with Tegafur after resection soon, and TACE in 4 or 8 weeks after resection.
  Interventions: Procedure: TACE+Tegafur
- TACE (Experimental): Patients will be treated with TACE alone in 4 or 8 weeks after resection.
  Interventions: Procedure: TACE

INTERVENTIONS:
Procedure: TACE+Tegafur — Tegafur: 40mg bid for 3 continuous months in 4 months. TACE: 4 or 8 weeks after resection.
  Other Names: TACE followed by Tegafur
  Arms: TACE+ Tegafur
Procedure: TACE — TACE alone
  Arms: TACE

SUMMARY:
The aim of this study is to compare the outcomes of Transarterial Chemoembolization (TACE) plus Tegafur with TACE alone in patients with intrahepatic cholangiocarcinoma after curative resection

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients > 18 years and <=70 years of age.
* Pathological evidence of ICC
* Tumors can be completely resected.
* Criteria of liver function: Child A-B level, serum bilirubin ≤ 1.5 times the upper limit of normal value, alanine aminotransferase and aspartate aminotransferase ≤ 2 times the upper limit of normal value.
* Patients who can understand this trial and have signed information consent.

Exclusion Criteria:

* Tumors can not be resected .
* Patients with apparent cardiac, pulmonary, cerebral and renal dysfunction, which may affect the treatment of Intrahepatic cholangiocarcinoma.
* Patients with a medical history of other malignant tumors.
* Subjects participating in other clinical trials.
* Liver function:Child C.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival rates of each group | 3 years

SECONDARY OUTCOMES:
Occurrence rate of recurrence of each group | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern hepatobilliary surgery hospital, Shanghai, Shanghai Municipality, China